CLINICAL TRIAL: NCT02071368
Title: A Single-Dose, Open-Label, Randomized, 3-Way Crossover Pivotal Study to Assess the Bioequivalence of the Fixed Dose Combination Tablets of Canagliflozin and Metformin Extended Release (XR) (2 x 150 mg/500 mg) With Respect to the Individual Components of Canagliflozin (1 x 300 mg) and Metformin XR Tablet (2 x 500 mg) in Healthy Fed Subjects
Brief Title: A Bioequivalence Study of the Fixed Dose Combination Tablets of Canagliflozin and Metformin Extended Release (XR) With Respect to the Individual Components in Healthy Fed Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR103258; 28431754DIA1063 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-02-24; First posted 2014-02-25 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Healthy; Canagliflozin; Metformin; JNJ-28431754; GLUMETZA®; Bioequivalence; Fixed Dose Combination
MeSH Terms: interventions — Canagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): Each participant will receive a single dose of 1 tablet of canagliflozin (CANA), 300 mg, and 2 tablets of metformin extended release (MET XR), 500 mg, administered together under fed conditions.
  Interventions: Drug: Canagliflozin, 300 mg; Drug: Metformin XR, 500 mg
- Treatment B (Experimental): Each participant will receive a single dose of 2 tablets of CANA/MET XR FDC (2 x [150 mg/500 mg]) formulation 1, under fed conditions.
  Interventions: Drug: CANA/MET XR FDC, Formulation 1, 150 mg/500
- Treatment C (Experimental): Each participant will receive a single dose of 2 tablets of CANA/MET XR FDC (2 x [150 mg/500 mg]), formulation 2, under fed conditions.
  Interventions: Drug: CANA/MET XR FDC, Formulation 2, 150 mg/500 mg

INTERVENTIONS:
Drug: Canagliflozin, 300 mg — Each tablet contains canagliflozin (CANA) of 300 mg to be taken orally (by mouth).
  Arms: Treatment A
Drug: Metformin XR, 500 mg — Each tablet contains metformin extended release (MET XR), 500 mg, to be taken orally (by mouth).
  Other Names: GLUMETZA
  Arms: Treatment A
Drug: CANA/MET XR FDC, Formulation 1, 150 mg/500 — Each tablet contains 150 mg of canagliflozin and 500 mg of metformin HCl granulate, formulation 1, to be taken orally.
  Arms: Treatment B
Drug: CANA/MET XR FDC, Formulation 2, 150 mg/500 mg — Each tablet contains 150 mg of canagliflozin and 500 mg of metformin HCl granulate, formulation 2, to be taken orally.
  Arms: Treatment C

SUMMARY:
The purpose of this study is to assess the bioequivalence (similarity of the drug amount in blood among the formulations) of the fixed dose combination (two components combined in one tablet) of canagliflozin and metformin extended release (XR) tablet (dose of 2 X 150 mg/500mg) with respect to the individual components of canagliflozin (1 x 300 mg) and metformin XR tablet (2 x 500 mg) in healthy fed participants.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), open-label (physicians and participants know the identity of the assigned treatment), single-center, single-dose, 3-treatment, 3-way crossover (the same medications provided to all participants but in different sequence) study of a Fixed Dose Combination (FDC) tablets of canagliflozin (CANA) and metformin extended release (MET XR) in comparison with tablets of individual components. Two FDC tablets will be studied with different formulations of MET XR component (CANA component will be identical). Both FDCs will be of the same strength: 2 tablets of 150mg CANA/500mg MET XR and will be compared with the equal doses of the individual drugs: canagliflozin (1 x 300mg tablet) and metformin XR (2 x 500mg tablets). Thus, there will be 3 treatment periods in the study: Treatment A: "Reference" treatment of individual components. Treatment B: CANA/MET XR FDC, formulation 1; and Treatment C: CANA/MET XR FDC, formulation 2. Approximately 42 healthy adult participants will be randomly assigned to 1 of 3 treatments groups, and then each group will receive all three treatments in different sequences (3-way crossover). The study will consist of 3 phases: a Screening Phase of approximately 3 weeks (Days -22 to -2), an Open-Label Treatment Phase consisting of 3 single-dose Treatment Periods of 5 days each (Days -1 through 4) separated by a washout of 10 to 14 days between Day 1 of each Treatment Period, and a Follow-up Phase occurring 7 to 10 days after the last study-related procedure on Day 4 of Treatment Period 3. The total duration of the study will be about 70 days for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent document indicating they understand the purpose of the study and procedures
* Must have a body mass index (BMI) of between 18 and 30 kg/m², inclusive
* Must have a body weight of not less than 50 kg
* Must have a blood pressure between 90 and 140 mmHg inclusive, systolic, and no higher than 90 mmHg diastolic at screening
* Must have normal renal function and no evidence of kidney damage (including abnormalities in blood or urine tests)

Exclusion Criteria:

* History of or current clinically significant medical illness
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements)
* History of clinically significant allergies, especially known hypersensitivity or intolerance to drugs or lactose
* Known allergy to heparin or history of heparin induced thrombocytopenia
* Donated blood or blood products or had substantial loss of blood within 3 months before screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of canagliflozin following the single dose of drug administration | Day 1 to Day 2 (predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours postdose); Day 3 (48 hour); and Day 4
  Plasma concentrations of canagliflozin are used to evaluate how long canagliflozin stays in the body.
Plasma concentration of metformin extended release following the single dose of drug administration | Day 1 to Day 2 (predose, 0.5, 1, 2, 4, 6, 8, 10, 12, 14, 16, 24, and 30 hours postdose); and Day 3 (36 hours)
  Plasma concentrations of metformin are used to evaluate how long it stays in the body.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to Day 10 of the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Tempe, Arizona, United States